CLINICAL TRIAL: NCT05551676
Title: Comparison of Lateral Parasagittal Approach and Transforaminal Epidural Approach in Lumbar Epidural Steroid Injection
Brief Title: Transforaminal and Parasagittal Approach in Lumbar Epidural Steroid Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Director, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lomber Epidural
Record Dates: First submitted 2022-08-29; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Lumbar Radiculopathy
Keywords: epidural steroid injection; transforaminal steroid injection; radicular pain
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transforaminal group (Active Comparator): Transforaminal steroid injection will be applied, 30 patients
  Interventions: Procedure: transforaminal group
- Lateral parasagittal group (Active Comparator): Lateral parasagittal steroid injection will be applied, 30 patients
  Interventions: Procedure: Lateral parasagittal group

INTERVENTIONS:
Procedure: transforaminal group — Epidural steroid injection will be applied with transforaminal approach accompanied by fluoroscopy.
  Arms: Transforaminal group
Procedure: Lateral parasagittal group — Epidural steroid injection will be applied with lateral parasagittal approach accompanied by scopy.
  Arms: Lateral parasagittal group

SUMMARY:
Lumbar epidural injection is used in the treatment of lumbar radicular pain. There are three different application methods: lateral parasagittal, midline interlaminar and transforaminal epidural injection. Investigator aimed to compare lateral parasagittal and transforaminal epidural injection methods. The purpose of the study is to determine which method is more efficient.

DETAILED DESCRIPTION:
It was planned to recruit 60 participants in the study. Interlaminar epidural steroid injection will be applied to 30 patients with midline and 30 patients with lateral parasagittal approach. All patients will receive Oswestry disability index before and 2-4-12 weeks after the procedure. All patients will receive Somatization Amplification Scale (SSAS) before the treatment. The results of the patients will be compared. It will be investigated which method is more effective.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral low back pain, radiculopathy

Exclusion Criteria:

* malignancy
* past back surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-06-22 (Estimated); Study Completion 2023-12-22 (Estimated)

PRIMARY OUTCOMES:
Oswestry disability index | baseline, week 4, week 12
  Oswestry Low Back Pain Disability Questionnaire, the Oswestry Disability Index helps to measure a patient's lower back pain. It evaluates the extent to which the patient's level of function is restricted by the pain, concentrating on the effects rather than the nature of the pain.
  0% to 20%: minimal disability 41%-60%: severe disability 61%-80%: crippled

OTHER OUTCOMES:
The SomatoSensory Amplification Scale | Baseline
  a 10-item self-report instrument designed to assess the tendency to detect somatic and visceral sensations and experience them as unusually intense, toxic and alarming.
  10: No symptom, 50: worst symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Taylan AKKAYA, Study Director — Diskapi TRH; Hüseyin Alp Alptekin, Study Chair — Diskapi TRH; Ezgi Can, Principal Investigator — Diskapi TRH
Locations (1):
- Diskapi Yildirim Beyazıt Teaching and Research Hospital, Ankara, Turkey (Türkiye)